CLINICAL TRIAL: NCT06057584
Title: The Neural Mechanism and Efficacy of Somatosensory Motor Integration Training on the Upper Extremity Somatosensory Motor Function in Patients With Chronic Stroke
Brief Title: Effect of Somatosensory Motor Intergration Training on Post-stroke Upper Limb Function.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202302039RINB
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Stroke
Keywords: stroke; somatosensory-motor integration; somatosensory; motor; randomized controlled trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- somatosensory-motor integration training (Experimental)
  Interventions: Behavioral: somatosensory-motor integration training
- pure somatosensory training (Active Comparator)
  Interventions: Behavioral: pure somatosensory training
- pure motor training (Active Comparator)
  Interventions: Behavioral: pure motor training

INTERVENTIONS:
Behavioral: somatosensory-motor integration training — Participants will use both hands to perform functional tasks requiring somatosensory discrimination to provide different somatosensory stimuli to facilitate motor control. The experimental group will receive somatosensory-motor integration training, 3-5 sessions a week, for a total of 15 sessions.
  Arms: somatosensory-motor integration training
Behavioral: pure somatosensory training — Participants will use the affected hand to perform somatosensory discrimination tasks, including limb position discrimination and object discrimination.The experimental group will receive pure somatosensory integration training, 3-5 sessions a week, for a total of 15 sessions.
  Arms: pure somatosensory training
Behavioral: pure motor training — Participants will conduct bilateral task-oriented training, but the training task does not require somatosensory discrimination. Each round only uses the same target and target position to repeatedly practice the functional task movements, but the target or target position is different in different rounds. The experimental group will receive pure motor integration training, 3-5 sessions a week, for a total of 15 sessions.
  Arms: pure motor training

SUMMARY:
Background: Most patients suffer from post-stroke somatosensory and motor impairments, and 50% to 70% of patients in the chronic stage still have upper extremity impairments that severely limit their functional independence and quality of life. Somatosensory and motor functions are closely related to each other. Previous evidence showed that somatosensory training or stimulation can modulate motor performance and enhance the efficacy of motor training, and motor training has the potential to promote the reorganization of the somatosensory cortex and enhance somatosensory-motor integration. Therefore, combining somatosensory and motor training may optimize the recovery of upper limb function. However, due to the small number of relevant empirical studies and the low quality of evidence, the effects and neural mechanisms of combined somatosensory and motor training compared with pure somatosensory training or pure motor training are still unknown or uncertain.

Purposes: This project will compare the immediate and long-term effects of somatosensory-motor integration training, pure motor training, and pure somatosensory training on the somatosensory and motor functions of patients with chronic stroke, and will investigate the neural mechanisms of somatosensory-motor recovery using neuroimaging and neurophysiological techniques.

Research methods: A single-blind (assessor-blinded) randomized controlled trial design will be used in this three-year project. A sample of 153 patients with chronic stroke will be recruited, and subjects who meet the selection criteria will undergo a baseline assessment and then be randomly assigned in stratified blocks to either the somatosensory-motor integration training group, pure somatosensory training group or pure motor training group. Subjects will receive three to five 60-minute sessions per week for a total of 15 sessions, followed by post-intervention (immediate effect) and three-month follow-up (long-term effect) assessments. Outcome measures will include neuroimaging (functional near-infrared spectroscopy.), and clinical scales (somatosensory function, motor function, upper extremity function, real life functional upper extremity performance., daily activities, and quality of life). The data will be analyzed using intention-to-treat analysis. The treatment effects within each group will be determined by paired t tests. The difference in effects among the three groups will be analyzed by analyses of covariate. Multiple linear regressions will also be used to explore the factors affecting the recovery of somatosensory and motor functions.

Expected results and contributions: The researchers expect that somatosensory-motor integration training, pure somatosensory training and pure motor training can all effectively improve the somatosensory and motor functions of patients with stroke. Among the three groups, somatosensory-motor integration training will show the greatest improvement in upper extremity function. The results of this project will provide empirical evidence on the effects and neural mechanisms of somatosensory-motor integration training, which will help clinicians select appropriate treatment strategies, facilitate clinical reasoning, and predict the recovery potential of somatosensory-motor function based on patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20.
2. Diagnosed with stroke.
3. Stroke duration ≥ 6 months.
4. Upper limb Brunnstrom stage III-V.
5. No severe muscle spasticity (Modified Ashworth Scale ≤ 2) in all segments of the affected upper limb.
6. Self-perceived or therapist-assessed somatosensory impairment.

Exclusion Criteria:

1. Significant cognitive impairment (Montreal Cognitive Assessment < 26).
2. Severe mental disorders (e.g., schizophrenia, major depression).
3. Substance abuse or alcoholism.
4. Claustrophobia.
5. Severe aphasia affecting comprehension and clear expression of somatosensory information.
6. Hemineglect.
7. Other muscle or joint problems affecting upper limb function (e.g., contractures, rheumatoid arthritis, myositis ossificans).
8. Concurrent participation in other somatosensory or motor therapy studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pre- and 3-month change in cerebral hemodynamics evaluated by functional near-infrared spectroscopy (fNIRS) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  fNIRS collects cerebral hemodynamic parameters in the bi-hemispheric sensory-motor cortices to estimate the changes in functional activation and functional connection of the corresponding brain areas before and after the intervention. The fNIRS system uses near-infrared light with two wavelengths of 760 nm and 850 nm, and 8 LED light sources and 8 sensors will be placed on the scalp of the sensory-action cortex of the left and right brain of the subject.
Pre- and 3-month change in functional ability of the upper extremities assessed by Action Research Arm Test (ARAT) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The ARAT is an operant test that assesses functional ability of the upper extremities. It includes grasping, holding, pinching, and gross motor. Higher scores represent better upper body functional capacity.
Pre- and 3-month change in motor function of the upper limbs assessed by Fugl-Meyer Assessment of Upper Extremity (FMA-UE) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The FMA-UE evaluates the motor function of the upper limbs. The higher the score, the better the motor function of the upper limbs.
Pre- and 3-month change in sensation assessed by Revised Nottingham Sensory Assessment (rNSA) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The rNSA evaluates the tactile sense of the face, trunk and upper and lower extremities. The tactile sense includes light touch, temperature, pinprick, pressure, tactile localization and sensory extinction. Stereognosis and proprioception will also be evaluated. Higher scores represent better somatosensory function.
Pre- and 3-month change in sensation assessed by Rivermead Assessment of Somatosensory Performance (RASP) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The RASP assesses sharp/dull discrimination, surface pressure touch, surface localization, temperature discrimination, sensory extinction, two-point discrimination, and proprioception. Higher scores represent better somatosensory function.

SECONDARY OUTCOMES:
Pre- and 3-month change in the frequency and movement quality in daily use of the affected upper limb assessed by Motor Activity Log (MAL) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The MAL evaluates the frequency and movement quality in daily use of the affected upper limb in patients with stroke or traumatic brain injury. The higher the score, the better the use frequency or movement quality of the affected upper limb.
Pre- and 3-month change in the performance, self-perceived difficulty, and ability of basic activities of daily living (ADL) assessed by The Barthel Index-based Supplementary Scales (BI-SS) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The BI-SS and BI comprehensively evaluate the performance, self-perceived difficulty, and ability of basic activities of daily living (ADL) . Higher scores represent better ADL performance, greater ADL ability, and simpler perceptions of ADL.
Pre- and 3-month change in the quality of life in patients assessed by Stroke Impact Scale 3.0 (ML-SIS) | Pre- and post-test (up to 5 weeks) and three-month follow-up
  The ML-SIS, a short version of the Stroke Impact Scale 3.0 based on machine learning methods, evaluates the quality of life in patients with stroke. It includes strength, memory, emotion, communication, activities of daily living, mobility, hand function and social participation. Higher scores represent better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan